CLINICAL TRIAL: NCT00455052
Title: A Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous XMT-1001 in Patients With Advanced Solid Tumors
Brief Title: A Study of Intravenous XMT-1001 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mersana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MER-001
Record Dates: First submitted 2007-04-01; First posted 2007-04-03 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-01

CONDITIONS: Small Cell Lung Cancer; Non-small Cell Lung Cancer
Keywords: XMT-1001; cancer; tumor; camptothecin; Fleximer; polymer; Phase 1; safety; pharmacokinetics; maximum tolerated dose; NSCLC; non-small cell lung cancer; SCLC; small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — XMT 1001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XMT-1001 (Experimental): XMT-1001 is administered I.V. every 21 days. Groups of 3 patients are given one dose and the dose increases for each group. The first dose level is 17 mg/m^2, the next dose level is 30 mg/m^2, followed by dose levels: 50 mg/m^2, 80 mg/m^2, 120 mg/m^2, 150 mg/m^2, and 190 mg/m^2 until disease progressions or unacceptable side effects are experienced.
  Interventions: Drug: XMT-1001

INTERVENTIONS:
Drug: XMT-1001 — XMT-1001 is administered as an IV infusion once every 21 days. This expansion of the Phase 1 study is to confirm the MTD.
  Other Names: MER-1001

SUMMARY:
This amended expansion phase of the protocol is to further the experience at a dose level of 150 mg CPT eq/m2 in patients with Stage IV non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC) and to test for preliminary anti-tumor activity in these tumor types. The MTD was initially defined as 113 mg CPT equivalents(eq)/m2 in the dose escalation part of the study. However, in the initial expansion phase (Protocol Amendment 11), 11 patients (10 NSCLC patients and 1 gastric cancer patients) were dosed at 113 mg CPT eq/m2 and less bone marrow toxicity was observed as compared to more heavily pre-treated patients in the dose escalation part of the study. Therefore, this amended expansion phase will investigate the safety and anti-tumor effects of a dose of 150 mg CPT eq/m2.

The study will also determine:

* The safety and tolerability of XMT-1001 at 150 mg CPT eq/m2
* The pharmacokinetics (PK) of XMT-1001 (how XMT-1001 behaves in the body) in patients Stage IV non-small cell lung carcinoma (NSCLC) and small cell lung cancer
* Evidence of XMT-1001 anti-tumor activity at 150 mg CPT eq/m2

DETAILED DESCRIPTION:
This is an open-label study of XMT-1001 administered intravenously over 4 hours every 21 days (1 Cycle). Blood sampling for PK analyses will be performed immediately prior to dosing, and 9 times after dosing. Patients will be assessed for toxicities known to occur with other drugs of this class, such as bone marrow suppression, elevated liver function enzymes, hemorrhagic cystitis, and diarrhea. Tumor imaging will be performed every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Have histological or cytological documentation of one of the following:

   A. NSCLC with Stage IV disease according to the American Joint Cancer Commission TNM Staging (7th Edition)
   * Have received at least one prior chemotherapy regimen but no more than two chemotherapy regimens for their advanced disease (not containing irinotecan or topotecan).
   * Adjuvant chemotherapy will be considered as a prior chemotherapy regimen only if it is completed less than 6 months prior to enrollment.
   * Treatment with erlotinib or crizotinib as single agents will not be considered as a chemotherapy regimen for purposes of this trial OR B. SCLC with Stage IV (extensive) or recurrent disease after definitive treatment for limited stage disease according to the American Joint Cancer Commission TNM Staging (7th Edition)1
   * Have received at least one prior chemotherapy regimen but no more than two chemotherapy regimens for their advanced disease (not containing irinotecan or topotecan).
   * Adjuvant chemotherapy will be considered as a prior chemotherapy regimen only if it is completed less than 6 months prior to enrollment.
3. Patients must be refractory or resistant to standard therapy or for whom standard therapy is not anticipated to be curative and who have progressed through prior regimens.
4. Patients must have measurable disease with at least one lesion that can be accurately measured by Response Evaluation Criteria in Solid Tumors (RECIST). The lesion size must be ≥20 mm by conventional radiological techniques or ≥10 mm by spiral CT scan. Disease in an irradiated field as the only site of measurable disease is acceptable if there has been a clear progression of the lesion. PET scans are not suitable for providing these measurements. For patients who are sensitive to contrast, MRI may be used.
5. Patients with CNS metastases are acceptable provided that the disease has been treated (e.g. surgery, whole brain radiotherapy, stereotactic radiotherapy etc.) and the patient is stable for at least two weeks and does not require steroids (at least one week off steroids). Anti-seizure medication is allowed at the discretion of the treating physician.
6. At least 42 days since administration of mitomycin or nitrosoureas, and 28 days since any other chemotherapy, investigational agent, and/or radiation therapy.
7. Have the following laboratory values:

   * Absolute neutrophil count (ANC) ≥1500 cells/mm3
   * Platelet count >100,000 cells/mm3
   * Hemoglobin ≥9.0 g/dL
   * Adequate renal function (serum creatinine ≤2 mg/dL) and creatinine clearance ≥45 mL/min (Calculated by Cockroft and Gault method)
   * Adequate hepatic function (bilirubin ≤1.5 mg/dL)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the institutional upper limit of normal (ULN, or

     * 5 times the ULN if liver metastases are present)
   * Albumin of >3.0 g/dL
   * PT and PTT ≤1.5 times the ULN
8. Have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1.
9. Have a life expectancy of at least 3 months.
10. Have signed an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Every 7 days in each 21 day cycle

SECONDARY OUTCOMES:
Tumor response | Every 2 cycles
Time to tumor progression | Every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Edward Sausville, MD, Principal Investigator — University of Maryland Greenebaum Cancer Center; Glen J Weiss, MD, Principal Investigator — TGen Clinical Research Services at Scottsdale Healthcare; Lawrence Garbo, MD, Principal Investigator — New York Oncology Hematology; Allen Lee Cohn, MD, Principal Investigator — Rocky Mountain Cancer Centers; Paul R. Conkling, MD, Principal Investigator — Virginia Oncology Associates; William J Edenfield, MD, Principal Investigator — Institute for Translational Oncology Research; Donald A. Richards, MD, Principal Investigator — Texas Oncology - Tyler; John R. Caton, MD, Principal Investigator — Willamette Valley Cancer Institute and Research Center; David A. Smith, MD, Principal Investigator — Northwest Cancer Specialists - Vancouver Cancer Center; Hillary H. Wu, MD, Principal Investigator — Central Indiana Cancer Centers; Fadi Braiteh, MD, Principal Investigator — Comprehensive Cancer Centers of Nevada; Stephen Anthony, MD, Principal Investigator — Evergreen Hematology & Oncology
Locations (12):
- United States (12):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, New York, New York
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Institute of Translational Oncology Research, Greenville, South Carolina
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Evergreen Hematology & Oncology, Spokane, Washington
  - Vancouver Cancer Center, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yurkovetskiy AV, Hiller A, Syed S, Yin M, Lu XM, Fischman AJ, Papisov MI. Synthesis of a macromolecular camptothecin conjugate with dual phase drug release. Mol Pharm. 2004 Sep-Oct;1(5):375-82. doi: 10.1021/mp0499306. PMID 16026008